CLINICAL TRIAL: NCT00149188
Title: A Phase IV, Multicentre, Open Label, Controlled Study to Assess the Ability of Patients With Acromegaly, or Their Partners, to Administer Somatuline Autogel.
Brief Title: Somatuline Autogel: Acromegaly Self/Partner Injection Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y-97-52030-150
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Acromegaly
Keywords: Growth Hormone
MeSH Terms: conditions — Acromegaly | interventions — lanreotide

INTERVENTIONS:
Drug: Lanreotide (Autogel formulation)

SUMMARY:
The purpose of this study is to allow patients with acromegaly, or their partners, to learn how to successfully inject Somatuline Autogel at home. Ability to perform unsupervised injections whilst maintaining adequate disease control will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have a clinical diagnosis of acromegaly
* The patient must have been tested and shown to have a GH level less than or equal to 10 micrograms/L within 28 days prior to the baseline visit
* The patient must be currently treated with Somatuline Autogel and have been stable on their current dose for at least 6 months immediately prior to screening
* The patient must be able to store study medication in a refrigerator in their own home

Exclusion Criteria:

* The patient has had pituitary surgery (adenomectomy) within 6 months prior to screening
* The patient has received pituitary radiotherapy within one year prior to screening
* The patient is likely to require pituitary surgery (adenomectomy) or to receive radiotherapy during the study period
* The patient is currently receiving a GH antagonist or a somatostatin analogue other than Somatuline Autogel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-02; Primary Completion 2005-08-24 (Actual); Study Completion 2005-08-24 (Actual)

PRIMARY OUTCOMES:
To assess the ability of patients or their partners to perform unsupervised Somatuline Autogel injections.

SECONDARY OUTCOMES:
To assess whether administration of unsupervised injections of Somatuline Autogel has any effect on GH and IGF-1 control or serum lanreotide levels.
To assess patient/partner and healthcare professional experience with unsupervised injections.
To assess the safety of patients or their partners performance of unsupervised Somatuline Autogel injections.

CONTACTS AND LOCATIONS:
Overall Officials: UK Medical Director, MD, Study Director — Ipsen
Locations (10):
- United Kingdom (10):
  - Michael White Centre Diabetes & Endocrinology, Hull Royal Infirmary, Hull, East Yorkshire
  - Department of Endocrinology, The Royal Free Hospital, Hampstead, London
  - Dept of Endocrinology, Aberdeen Royal Infirmary, Aberdeen
  - Department of Medicine, Queen Elizabeth Hospital, Birmingham
  - Department of Endocrinology, Coventry & Warwickshire Hospital, Coventry
  - Department of Endocrinology, Leicester Royal Infirmary, Leicester
  - Department of Endocrinology, Manchester Royal Infirmary, Manchester
  - The Oxford Centre for Diabetes, Endocrinology and Metabolism, The Churcill Hospital, Oxford
  - Department of Endocrinology, Royal Hallamshire Hospital, Sheffield
  - Department of Endocrinology, Sunderland Royal Hospital, Sunderland

REFERENCES:
- [Result] Bevan JS, Newell-Price J, Wass JA, Atkin SL, Bouloux PM, Chapman J, Davis JR, Howlett TA, Randeva HS, Stewart PM, Viswanath A. Home administration of lanreotide Autogel by patients with acromegaly, or their partners, is safe and effective. Clin Endocrinol (Oxf). 2008 Mar;68(3):343-9. doi: 10.1111/j.1365-2265.2007.03044.x. Epub 2007 Sep 24. PMID 17892497